CLINICAL TRIAL: NCT02235064
Title: Prophylactic Use of Immediate Postpartum Sertraline to Prevent Postpartum Depression: A Double Blind Randomized Placebo Controlled Trial
Brief Title: Prophylactic Use of Postpartum Sertraline to Prevent Postpartum Depression
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low recruitment, completion of funding cycle
Sponsor: The Cooper Health System (Other)
Responsible Party: Principal Investigator, Richard Fischer MD, Professor, Department of OB/GYN, Cooper Medical School of Rowan University, The Cooper Health System
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CUH IRB#: 14-078
Record Dates: First submitted 2014-08-08; First posted 2014-09-09 (Estimated); Results first posted 2017-04-10 (Actual); Last update posted 2018-03-29 (Actual); Status verified 2018-02

CONDITIONS: Depression, Postpartum
MeSH Terms: conditions — Depression, Postpartum | interventions — Sertraline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sertraline (Experimental): Capsules containing crushed sertraline 50 mg combined with identically colored cellulose, daily for 12 weeks, followed by 4 day 25 mg taper
  Interventions: Drug: Sertraline
- Placebo (Placebo Comparator): Identical appearing capsule daily containing color-matched cellulose only
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sertraline — Capsule containing crushed sertraline 50 mg tablets mixed with identically colored cellulose, with 4 day 25 mg taper
  Other Names: Zoloft
  Arms: Sertraline
Drug: Placebo — Capsule containing cellulose powder of same color as experimental arm
  Other Names: Cellulose powder
  Arms: Placebo

SUMMARY:
The purpose of this project is to assess the effectiveness of preventative antidepressants immediately following delivery on postpartum depression rates in women at high risk due to prior history of depression or postpartum depression.

DETAILED DESCRIPTION:
Eligible women for our study would be identified antepartum from our three obstetrical groups delivering at Cooper University Hospital: Cooper Faculty Group, Women's Care Center, and CamCare. Potentially eligible women would be referred to the study coordinator or principal investigator to discuss the nature of the study. Those women who agreed to the trial would be further screened with a baseline structured psychiatric evaluation in the third trimester of the pregnancy to rule-out current depressive illness. If there was no evidence of depression at the antepartum evaluation, patients delivering a liveborn singleton fetus at 34 0/7 weeks or greater would be re-evaluated prior to discharge and, if scoring </= 12 on the Edinburgh Postpartum Depression scale, would then be enrolled in the trial.

Patients would be assigned to either sertraline 50 mg daily or identical appearing placebo for 12 weeks. Group allocation would be determined by restricted-randomization technique with variable block length, with the sequence generated by someone not associated with participant assignment. Assignment would be kept in sequentially numbered, opaque, sealed envelopes (SNOSE) in the pharmacy, which would dispense the medication (or placebo). Patients would be given a 30 day supply on the day of discharge, with refills provided by the study coordinator (through the pharmacy)for 12 weeks and a four-day supply of 25 mg Sertraline or placebo at the end of 12 weeks as a taper. Patients would also undergo follow-up blinded structured psychiatric evaluations at 4 weeks, 8 weeks, and 12 weeks to assess for adverse reaction to the assigned treatment agent, and for administration of questionnaires/evaluation to assess for development of depression. Any patient with recognized clinical depression would immediately be removed from further active participation in the study and referred to our Cooper Psychiatry department or outside psychiatrist for ongoing evaluation and treatment. Medication received (Sertraline or Placebo) would necessarily be revealed to Psych only for purposes of guiding appropriate further treatment.

All women randomized would be analyzed according to group assignment (intent-to-treat). Demographic information, including patient age, race/ethnicity, gravidity, parity, gestational age at delivery, infant birth weight, as well as infant weights from standard Pediatric visits (obtained verbally from the mother)would be recorded and compared using the Student t-test for normally distributed continuous data, Mann-Whitney U for non-normative continuous data, and the Chi Square test or Fisher Exact test for categorical data.

A sample size calculation was performed. Based on an anticipated rate of postpartum depression (PPD) of 30% in the placebo group, we would need 62 subjects in each group to detect a reduction in PPD to 10% in the sertraline group, with a power of .8 and a Type I error of .05. Based on the 2200 deliveries occurring annually at Cooper University Hospital, we anticipate that it would take 2-3 years to recruit 124 subjects into this study.

ELIGIBILITY:
Inclusion Criteria:

1. Past history of depression or postpartum depression
2. Singleton gestation
3. Delivery > 34 weeks gestation
4. No current clinical evidence of depression
5. Able to read and understand written English language

Exclusion Criteria:

1. Multiple gestation
2. Delivery prior to 34 weeks
3. Delivery outside of Cooper University Hospital
4. Major fetal anomaly or fetal demise
5. Current use of antidepressants
6. Evidence of active depression at antepartum evaluation
7. Edinburgh Postpartum Depression scale of >12 prior to discharge from the hospital
8. Maternal age < 18 years
9. Infant in Neonatal Intensive Care Unit (NICU) at time of patient discharge from hospital
10. Known or suspected allergy to Sertraline

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2014-07; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard L Fischer, M.D., Principal Investigator — Cooper Health System
Locations (1):
- Cooper University Hospital, Camden, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No
Only aggregate data to be reported

REFERENCES:
- [Background] Chambers CD, Hernandez-Diaz S, Van Marter LJ, Werler MM, Louik C, Jones KL, Mitchell AA. Selective serotonin-reuptake inhibitors and risk of persistent pulmonary hypertension of the newborn. N Engl J Med. 2006 Feb 9;354(6):579-87. doi: 10.1056/NEJMoa052744. PMID 16467545
- [Background] Gold LH. Postpartum disorders in primary care: diagnosis and treatment. Prim Care. 2002 Mar;29(1):27-41, vi. doi: 10.1016/s0095-4543(03)00072-1. PMID 11856657
- [Background] ACOG Committee on Practice Bulletins--Obstetrics. ACOG Practice Bulletin: Clinical management guidelines for obstetrician-gynecologists number 92, April 2008 (replaces practice bulletin number 87, November 2007). Use of psychiatric medications during pregnancy and lactation. Obstet Gynecol. 2008 Apr;111(4):1001-20. doi: 10.1097/AOG.0b013e31816fd910. No abstract available. PMID 18378767
- [Background] Howard LM, Hoffbrand S, Henshaw C, Boath L, Bradley E. Antidepressant prevention of postnatal depression. Cochrane Database Syst Rev. 2005 Apr 18;(2):CD004363. doi: 10.1002/14651858.CD004363.pub2. PMID 15846711
- [Background] Malm H, Klaukka T, Neuvonen PJ. Risks associated with selective serotonin reuptake inhibitors in pregnancy. Obstet Gynecol. 2005 Dec;106(6):1289-96. doi: 10.1097/01.AOG.0000187302.61812.53. PMID 16319254
- [Background] Moses-Kolko EL, Bogen D, Perel J, Bregar A, Uhl K, Levin B, Wisner KL. Neonatal signs after late in utero exposure to serotonin reuptake inhibitors: literature review and implications for clinical applications. JAMA. 2005 May 18;293(19):2372-83. doi: 10.1001/jama.293.19.2372. PMID 15900008
- [Background] Payne JL. Antidepressant use in the postpartum period: practical considerations. Am J Psychiatry. 2007 Sep;164(9):1329-32. doi: 10.1176/appi.ajp.2007.07030390. No abstract available. PMID 17728416
- [Background] Pearlstein T, Howard M, Salisbury A, Zlotnick C. Postpartum depression. Am J Obstet Gynecol. 2009 Apr;200(4):357-64. doi: 10.1016/j.ajog.2008.11.033. PMID 19318144
- [Background] Safety of SSRIs in Pregnancy. Med Lett Drugs Ther. 2008 Nov 17;50(1299):89-91. No abstract available. PMID 19008787
- [Background] Sanz EJ, De-las-Cuevas C, Kiuru A, Bate A, Edwards R. Selective serotonin reuptake inhibitors in pregnant women and neonatal withdrawal syndrome: a database analysis. Lancet. 2005 Feb 5-11;365(9458):482-7. doi: 10.1016/S0140-6736(05)17865-9. PMID 15705457
- [Background] Wisner KL, Perel JM, Peindl KS, Hanusa BH, Piontek CM, Findling RL. Prevention of postpartum depression: a pilot randomized clinical trial. Am J Psychiatry. 2004 Jul;161(7):1290-2. doi: 10.1176/appi.ajp.161.7.1290. PMID 15229064
- [Background] Wisner KL, Perel JM, Peindl KS, Hanusa BH, Findling RL, Rapport D. Prevention of recurrent postpartum depression: a randomized clinical trial. J Clin Psychiatry. 2001 Feb;62(2):82-6. doi: 10.4088/jcp.v62n0202. PMID 11247106
- [Background] Yonkers KA, Wisner KL, Stewart DE, Oberlander TF, Dell DL, Stotland N, Ramin S, Chaudron L, Lockwood C. The management of depression during pregnancy: a report from the American Psychiatric Association and the American College of Obstetricians and Gynecologists. Obstet Gynecol. 2009 Sep;114(3):703-713. doi: 10.1097/AOG.0b013e3181ba0632. PMID 19701065

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Sertraline | Placebo
Started | 1 | 1
Completed | 1 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sertraline | Placebo | Total
Number analyzed (Participants) | 1 | 1 | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 1 | 2
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 33 [33 to 33] | 30 [30 to 30] | 31.5 [30 to 33]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Development of Postpartum Depression up to 12 Weeks Following Discharge From Hospital
Description: Patients met with single psychiatrist (co-investigator), blinded to group assignment, who evaluated the patient using Edinburgh Postpartum Depression Screen, Hamilton Depression Rating Scale, Global Assessment of Functioning Scale, and clinical assessment
  0 = No postpartum depression up to 12 weeks following discharge from hospital
  1 = Postpartum depression up to 12 weeks following discharge from hospital
Time Frame: Discharge from hospital to 12 weeks postpartum
Measure: Count of Participants; unit: Participants
Arm/Group | Sertraline | Placebo
Number analyzed (Participants) | 1 | 1
Participants | 0 | 0

2. Secondary Outcome: Number of Participants With Adverse Reaction to Treatment Agent up to 12 Weeks Following Discharge From Hospital
Description: The Antidepressant Side-Effect Checklist (ASEC) was employed to detect any adverse reaction to treatment regimens
Time Frame: Discharge from hospital to 12 weeks postpartum
Measure: Count of Participants; unit: Participants
Arm/Group | Sertraline | Placebo
Number analyzed (Participants) | 1 | 1
Participants | 0 | 1

3. Secondary Outcome: Reported Infant Weight at 4 Weeks Following Delivery
Time Frame: 4 weeks postpartum
Measure: Mean (Full Range); unit: Grams
Arm/Group | Sertraline | Placebo
Number analyzed (Participants) | 1 | 1
Grams | 3033 [3033 to 3033] | 2750 [2750 to 2750]

4. Secondary Outcome: Number of Participants With Perceived Infant Sleeping Difficulty at 4 Weeks Postpartum
Time Frame: 4 weeks postpartum
Measure: Count of Participants; unit: Participants
Arm/Group | Sertraline | Placebo
Number analyzed (Participants) | 1 | 1
Participants | 0 | 0

5. Secondary Outcome: Number of Participants With Perceived Infant Feeding Difficulties 4 Weeks Postpartum
Time Frame: 4 weeks postpartum
Measure: Count of Participants; unit: Participants
Arm/Group | Sertraline | Placebo
Number analyzed (Participants) | 1 | 1
Participants | 0 | 0

6. Secondary Outcome: Reported Infant Weight at 8 Weeks Following Delivery
Time Frame: 8 weeks postpartum
Measure: Mean (Full Range); unit: Grams
Arm/Group | Sertraline | Placebo
Number analyzed (Participants) | 1 | 1
Grams | 5301 [5301 to 5301] | 3685 [3685 to 3685]

7. Secondary Outcome: Reported Infant Weight at 12 Weeks Following Delivery
Time Frame: 12 weeks postpartum
Measure: Mean (Full Range); unit: Grams
Arm/Group | Sertraline | Placebo
Number analyzed (Participants) | 1 | 1
Grams | 5301 [5301 to 5301] | 4734 [4734 to 4734]

8. Secondary Outcome: Number of Participants With Perceived Infant Sleeping Difficulty at 8 Weeks Postpartum
Time Frame: 8 weeks postpartum
Measure: Count of Participants; unit: Participants
Arm/Group | Sertraline | Placebo
Number analyzed (Participants) | 1 | 1
Participants | 0 | 0

9. Secondary Outcome: Number of Participants With Perceived Infant Sleeping Difficulty at 12 Weeks Postpartum
Time Frame: 12 weeks postpartum
Measure: Count of Participants; unit: Participants
Arm/Group | Sertraline | Placebo
Number analyzed (Participants) | 1 | 1
Participants | 0 | 0

10. Secondary Outcome: Number of Participants With Perceived Infant Feeding Difficulties 8 Weeks Postpartum
Time Frame: 8 weeks postpartum
Measure: Count of Participants; unit: Participants
Arm/Group | Sertraline | Placebo
Number analyzed (Participants) | 1 | 1
Participants | 0 | 0

11. Secondary Outcome: Number of Participants With Perceived Infant Feeding Difficulties 12 Weeks Postpartum
Time Frame: 12 weeks postpartum
Measure: Count of Participants; unit: Participants
Arm/Group | Sertraline | Placebo
Number analyzed (Participants) | 1 | 1
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Sertraline | Placebo
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/1
Other Adverse Events (participants affected / at risk) | 0/1 | 1/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sertraline (N=1) | Placebo (N=1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes